CLINICAL TRIAL: NCT02449616
Title: Evaluation of Repeat Administration of Purified Poloxamer 188 in Vaso-Occlusive Crisis of Sickle Cell Disease (EPIC-E): An Open-Label Safety Extension Trial Assessing Repeat Administration of MST-188 (Purified Poloxamer 188) Injection in Subjects With Sickle Cell Disease Experiencing Vaso Occlusive Crisis
Brief Title: Evaluation of Repeat Administration of Purified Poloxamer 188
Acronym: EPIC-E
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mast Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MST-188-04
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell; vaso-occlusive crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Drug (Experimental): MST-188
  Interventions: Drug: MST-188

INTERVENTIONS:
Drug: MST-188 — Intravenous administration as 100 mg/kg for 1 hour followed by 30 mg/kg/hour for up to 48 hours.
  Other Names: vepoloxamer

SUMMARY:
The purpose of this study is to evaluate the safety of repeat administration of MST-188 during vaso-occlusive crisis of sickle cell disease. Additionally, this study will evaluate the development of acute chest syndrome during VOC and re-hospitalization for recurrence of VOC.

ELIGIBILITY:
Inclusion Criteria:

* Completed participation in study MST-188-01 (EPIC study)
* Subject age 4 through 65 years
* Subject is experiencing acute pain typical of VOC and requires treatment with parenteral opioid analgesia
* Subject requires hospitalization

Exclusion Criteria:

* Subject has acute chest syndrome
* Subject's laboratory results indicate inadequate organ function
* Subject is pregnant or nursing an infant
* Subject had a painful crisis requiring hospitalization within the preceding 14 days
* Subject has been transfused within the past 14 days
* Subject has complications related to SCD

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Safety as measured as the incidence of adverse events | 30 days after administration of study drug

SECONDARY OUTCOMES:
Rate of re-hospitalization for recurrence of VOC | Within 14 days of the date of discharge
Occurrence of acute chest syndrome | Within 120 hours of registration

CONTACTS AND LOCATIONS:
Overall Officials: Edwin L Parsley, D. O., Study Director — Mast Therapeutics, Inc.
Locations (9):
- United States (9):
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Joe Dimaggio Children's Hospital, Hollywood, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Our Lady of the Lake Children's Hospital, Baton Rouge, Louisiana
  - Rutgers University, New Brunswick, New Jersey
  - Medical University of South Carolina, Charleston, South Carolina
  - T. C. Thompson Children's Hospital, Chattanooga, Tennessee